CLINICAL TRIAL: NCT05398406
Title: Subcostal Transversus Abdominus Plane Block, Erector Spinae Plane Block and Paravertebral Blocks Effects
Brief Title: Subcostal Transversus Abdominus , Erector Spinae and Paravertebral Blocks Effects on Laparoscopic Cholecystectomy Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Arzu Esen Tekeli, Associate Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 01
Record Dates: First submitted 2022-05-17; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Comparison; Evaluation
Keywords: plane blocks; ultrasonography; bupivacaine

STUDY DESIGN:
Intervention Model Description: randomized, single-blind, closed-envelope method
Who Masked: Participant
Masking Description: Cases; under the age of 20 - over 60, emerge and bleeding, outside the ASAI-II functional status, undergo surgery other than laparoscopic cholecystectomy, refused to participate in the study, allergic to local anesthetic agents, with a body mass index (BMI) >30, have contraindications for regional anesthesia (sepsis, local infection, coagulopathy, heart disease, hypovolemia, cases that do not want regional anesthesia), pregnant were not included in the study.Twenty patients in each group and a total of 60 patients were included the study by power analysis. According to the randomized, single-blind, closed-envelope method, patients were randomly divided into three groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subcostal TAP Block (Experimental): In the supine position, the US probe was placed on the imaginary line connecting the anterior superior iliac spine (SIAS) and the umbilicus. The ilioinguinal and iliohypogastric nerves in the fascia of the internal obliq and transverse abdominis muscles were visualized by US. A total of 40 ml (20+20 ml) of local anesthetic was infiltrated around the nerve bilaterally with a 100 mm 21G peripheral nerve block needle (SonoPlex Stim Cannula, PAJUNK®,USA).
  Interventions: Other: TAP Block group
- ESP Block (Experimental): In the lateral decubitus position, a 100 mm 21G peripheral nerve block needle (SonoPlex Stim Cannula, PAJUNK®,USA) was inserted between the erector spinae muscle and the transverse process structures in an in-plane section guided by US from the T7-8 level. A total of 40 ml of the prepared solutions were injected bilaterally as 20+20 ml.
  Interventions: Other: Erector spinae block group
- Paravertebral block (Experimental): In the lateral decubitus position, the cranial to caudal transverse processes and the superior costotransverse ligament and the pleura were visualized from the T7-8 level in the in-plane section under US guidance. A 100 mm 21G peripheral nerve block needle (SonoPlex Stim Cannula, PAJUNK®, USA) was advanced until it passed through the superior costotransverse ligament. A total of 40 ml of injections were made bilaterally in the form of 20+20 ml.
  Interventions: Other: Paravertebral block group

INTERVENTIONS:
Other: TAP Block group — TAP Block: the US probe was placed on the imaginary line connecting the anterior superior iliac spine and the umbilicus. The ilioinguinal and iliohypogastric nerves in the fascia of the internal obliq and transverse abdominis muscles were visualized by US. A total of 40 ml of local anesthetic was infiltrated ESP Blok : a 100 mm 21G peripheral nerve block needle was inserted between the erector spinae muscle and the transverse process structures in an in-plane section guided by US from the T7-8 level. 40 ml of the prepared solutions were injected PVB: In the lateral decubitus position, the cranial to caudal transverse processes and the superior costotransverse ligament and the pleura were visualized from the T7-8 level in the in-plane section under US guidance. A 100 mm 21G peripheral nerve block needle was advanced until it passed through the superior costotransverse ligament. A total of 40 ml of injections were made
  Other Names: Paravertebral block group; Erector spinae block group
  Arms: Subcostal TAP Block
Other: Paravertebral block group — In the lateral decubitus position, the cranial to caudal transverse processes and the superior costotransverse ligament and the pleura were visualized from the T7-8 level in the in-plane section under US guidance. A 100 mm 21G peripheral nerve block needle (SonoPlex Stim Cannula, PAJUNK®, USA) was advanced until it passed through the superior costotransverse ligament. A total of 40 ml of injections were made bilaterally in the form of 20+20 ml.
  Other Names: PVB group
  Arms: Paravertebral block
Other: Erector spinae block group — In the lateral decubitus position, a 100 mm 21G peripheral nerve block needle (SonoPlex Stim Cannula, PAJUNK®,USA) was inserted between the erector spinae muscle and the transverse process structures in an in-plane section guided by US from the T7-8 level. A total of 40 ml of the prepared solutions were injected bilaterally as 20+20 ml.
  Other Names: ESP block group
  Arms: ESP Block

SUMMARY:
Sixty patients with ASA (American Society of Anesthesiologist) I-II physical status between the ages of 20-60 were randomized into three groups: TAP block group (Group T), ESP block group (Group E) and PVB group (Group P). Bilateral 20cc (total 40cc for each patient) 0.25% bupivacaine was applied by ultrasound (US) guidance. Intraoperative vital signs (heart rate, blood pressure, and saturation), Train-of-four (TOF) values, additional dose of opioid and muscle relaxant needs, complications were recorded. Postoperative side effects (nausea, vomiting, itching, tremor), the need for additional postoperative analgesia, Visual Analog Scale (VAS) scores were noted.

DETAILED DESCRIPTION:
Cases; under the age of 20 - over 60, emerge and bleeding, outside the ASAI-II functional status, undergo surgery other than laparoscopic cholecystectomy, refused to participate in the study, allergic to local anesthetic agents, with a body mass index (BMI) >30, have contraindications for regional anesthesia (sepsis, local infection, coagulopathy, heart disease, hypovolemia, cases that do not want regional anesthesia), pregnant were not included in the study.Twenty patients in each group and a total of 60 patients were included the study by power analysis. According to the randomized, single-blind, closed-envelope method, patients were randomly divided into three groups.

Group T (Subcostal TAP Block): 40 cc (20cc+20cc) 0.25 % Bupivacaine for bilateral application Group E (ESP Block): 40 cc (20cc+20cc) 0.25% Bupivacaine for bilateral application Group P (PVB): 40 cc (20cc+20cc) 0.25% Bupivacaine for bilateral application were prepared.

ELIGIBILITY:
Inclusion Criteria:

* 20-60 years,
* ASA I-II ,
* scheduled for elective laparoscopic cholecystectomy
* under general anesthesia,
* agreed to participate in the study,

Exclusion Criteria:

* under the age of 20 - over 60,
* emerge and bleeding,
* outside the ASAI-II functional status,
* undergo surgery other than laparoscopic cholecystectomy,
* refused to participate in the study, allergic to local anesthetic agents,
* body mass index (BMI) >30,
* have contraindications for regional anesthesia (sepsis, local infection, coagulopathy, heart disease, hypovolemia, cases that do not want regional anesthesia),
* pregnant

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
demographic data | 6 monthes
  age, gender, height, weight, and BMI
Heart rate values | 6 monthes
  Heart rate values for (-5)-0-30-40 min

SECONDARY OUTCOMES:
postoperative analgesic requirement | 6 monthes
  the need for postoperative analgesia
postoperative side effects | 6 monthes
  nausea, vomiting and tremor

CONTACTS AND LOCATIONS:
Overall Officials: Arzu E Tekeli, MD, Principal Investigator — Yuzuncu Yil University
Locations (1):
- Van Yuzuncu Yil University, Van, Tuşba, Turkey (Türkiye)